CLINICAL TRIAL: NCT04572789
Title: Omega-3 Fatty Acid in the Prevention of Migraine: From the Randomized Clinical Trial to Molecular Biology Approaches
Brief Title: Omega-3 Fatty Acid in the Prevention of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Chun-pai Yang, MD, Director, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10844
Record Dates: First submitted 2020-09-23; First posted 2020-10-01 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Migraine; Omega-3 Polyunsaturated Fatty Acids
MeSH Terms: conditions — Migraine Disorders | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-6

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): All participants will complete a set of outcome measures at baseline and the follow-up visits before and after 12 weeks of placebo omega-6 PUFAs intervention and a series of blood tests for neurotransmitter, neurotrophic and neuroinflammation. The clinical efficacy and the peripheral blood biomarkers, will be analyzed at baseline and the end of the intervention.
  Interventions: Dietary Supplement: omega-6 PUFAs
- Omega-3 (Experimental): All participants will complete a set of outcome measures at baseline and the follow-up visits before and after 12 weeks of omega-3 PUFAs intervention (EPA) and a series of blood tests for neurotransmitter, neurotrophic and neuroinflammation. The clinical efficacy and the peripheral blood biomarkers, will be analyzed at baseline and the end of the intervention.
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acids — All participants will complete a set of outcome measures at baseline and the follow-up visits before and after 12 weeks of omega-3 PUFAs intervention (EPA, 1.8 g/day) and a series of blood tests for neurotransmitter, neurotrophic and neuroinflammation. The clinical efficacy and the peripheral blood biomarkers, will be analyzed at baseline and the end of the intervention.
  Arms: Omega-3
Dietary Supplement: omega-6 PUFAs — All participants will complete a set of outcome measures at baseline and the follow-up visits before and after 12 weeks of placebo omega-6 PUFAs intervention and a series of blood tests for neurotransmitter, neurotrophic and neuroinflammation. The clinical efficacy and the peripheral blood biomarkers, will be analyzed at baseline and the end of the intervention.
  Arms: placebo

SUMMARY:
To understand the clinical efficacy for omega-3 PUFAs migraine prevention.To uncover the underlying biochemical or neurophysiological mechanisms by which omega-3 PUFAs for migraine prevention.

DETAILED DESCRIPTION:
Background:

Migraine is a common disabling disorder and its substantial burden is associated with considerable negative impact on quality of life. Several pharmacological treatments are available for migraine prophylaxis but insufficient efficacy and significant side effects preclude their widely use for migraine treatment. In recent years, more attention has been paid to dietary supplements and natural ingredients for the treatment of migraine. Omega-3 polyunsaturated fatty acids (omega-3 PUFAs) have beneficial on the reduction of neurogenic, perivascular inflammations and pro-inflammatory cytokines, which may play an important role in the pathophysiology of migraine. However, the results of investigations carried out about the clinical efficacy of omega-3 PUFAs in the management of migraine are inconsistent.

Purpose:

To understand the clinical efficacy for omega-3 PUFAs migraine prevention. To uncover the underlying biochemical or neurophysiological mechanisms by which omega-3 PUFAs for migraine prevention

Method:

This two-year project includes clinical approaches to investigate the therapeutic effects of omega-3 PUFAs on episodic migraine (4-14 days/month) without migraine preventive treatment in the past one month. 120 patients, aged 20-65, will be randomized in a 12-week, double-blind, placebo-controlled trial comparing the effects of high-dose eicosapentaenoic acid (EPA, 1.8g/day) and placebo intervention. All participants will complete a set of outcome measures: headache questionnaires and headache diary, the Migraine Disability Assessment (MIDAS), patient overall impression questionnaire-migraine improvement questionnaire (PGI-I), patient overall impression questionnaire-migraine severity questionnaire (PGI-S), Beck Depression Inventory-II (BDI-II), Hospital anxiety and depression scale (HADS), Migraine Quality of Life Questionnaire (MSQ), Pittsburgh Sleep Quality Questionnaire (PSQI) at baseline and the follow-up visits before and after 12 weeks of placebo or omega-3 PUFAs intervention (EPA, 1.8 g/day) and a series of blood tests for neurotransmitter, neurotrophic and neuroinflammation. The clinical efficacy and the peripheral blood biomarkers, will be analyzed at baseline and the end of the intervention.

Expected results:

To establish the clinical evidence of omega-3 PUFAs on migraine prevention. To provide significant insights into molecular actions of omega-3 PUFAs on migraine prevention.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Aged 20 to 65 years old
   2. A diagnosis based on the International Classification of Headache Disorders (ICHD-3)
   3. An established migraine history for at least 1 year
   4. Independent from the study
   5. Written informed consent
2. Exclusion Criteria:

   1. Chronic migraine
   2. Headaches other than migraine
   3. Use any of the following drugs in the past four weeks：

      * Migraine prophylaxis agents
      * Anti-depressants
      * Calcium channel blockers
      * Anti-epileptic agents
      * Cycle-modulating hormonal drugs
      * Onabotulinumtoxin A (Botox) injection
   4. Migraine onset after the age of 50
   5. Emerging abnormal findings on：

      * Laboratory parameters
      * Physical examination
      * Suicidal risks
      * Severe depression
   6. Cognitive impairment
   7. Allergies or hypersensitivity to fish or omega-3 fatty acids
   8. Bleeding diathesis or using anticoagulation agents
   9. Pregnancy or nursing

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Reduction of migraine attacks during the 12-week period [Efficacy] | 12 weeks
  The primary end point is the mean change from baseline (28-day pretreatment period) in the mean number of monthly migraine days during the 12-week period. A migraine day was defined as (a day with headache pain that lasted 4 hours with a peak severity of moderate or severe intensity, or any severity or duration if the participant took and responded to a triptan or ergot) from the second to the fourth diaries compared with the first diary (baseline period).

SECONDARY OUTCOMES:
50% reduction of migraine attacks | 12 weeks
  50% reduction in the the average migraine attacks per month during the 12-week period from baseline (28-day pretreatment period).
Migraine Disability Assessment Score (MIDAS) | 12 weeks
  Change of MIDAS scores from baseline to endpoint.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Change of HADS scores from baseline to endpoint.
The Patient Global Impression of Improvement (PGI-I) and Patient Global Impression of Severity (PGI-S) | 12 weeks
  Change of PGI-I and PGI-S scores from baseline to endpoint.
The Beck Depression Inventory-II (BDI-II) | 12 weeks
  Change of BDI-II scores from baseline to endpoint.
Reduction of acute headache medications | 12 weeks
  Reduction from baseline in the number of days with acute headache medications, from the second to the fourth diaries compared with the first diary (baseline period).
Reduction of accumulative headache hours | 12 weeks
  Reduction in accumulative headache hours from the second to the fourth diaries compared with the first diary (baseline period).
Migraine Quality of Life Questionnaire (MSQ) scores | 12 weeks
  Change of Migraine Quality of Life Questionnaire (MSQ) scores from baseline to endpoint.
Pittsburgh Sleep Quality Questionnaire (PSQI) scores | 12 weeks
  Change of Pittsburgh Sleep Quality Questionnaire (PSQI) scores from baseline to endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pai Yang, Dr., Principal Investigator — Neurology department of Kuang Tien General hospital
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No